CLINICAL TRIAL: NCT01429207
Title: Phase I Study: Monitoring Levodopa-Induced Dyskinesia Using Accelerometer & Gyroscope-based Motion Detection System
Brief Title: Capturing Parkinson's Disease Medication Side Effects During Daily Activities
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 1R43NS071882-01A1 (NIH)
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson's Disease; Dyskinesia
Keywords: levodopa; tremor; bradykinesia; motion sensors
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Tremor; Hypokinesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of the study is to test whether body-worn wireless motion sensors can measure dyskinesias (involuntary movements caused by medications) in individuals with Parkinson disease (PD) independent of voluntary activity being performed and other PD motor symptoms (e.g. tremor).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable or definite idiopathic Parkinson Disease with motor fluctuations that include dyskinesias after taking their usual dose of levodopa/carbidopa

Exclusion Criteria:

* Antipsychotic medications (including quetiapine and clozapine)
* Coexisting neurologic disease such as stroke or dementia
* Lacking capacity for informed consent
* Residing in a nursing home
* comorbid non-neurologic illnesses that impacts the ability to perform the study tasks
* Implantable defibrillators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic PD demonstrating levodopa-induced dyskinesias
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-08

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States